CLINICAL TRIAL: NCT04202978
Title: Camrelizumab Combined With Apatinib 、XELOX 、RFA in the Treatment of Liver Metastases of Colorectal Cancer: One-arm Exploratory Clinical Study
Brief Title: Camrelizumab Combined With Apatinib 、XELOX 、RFA in the Treatment of Liver Metastases of Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-R002
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-02

CONDITIONS: Hepatic Metastasis of Colorectal Cancer
MeSH Terms: interventions — camrelizumab; apatinib; Capecitabine; Oxaliplatin; Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+ Apatinib +XELOX +RFA (Experimental): Camrelizumab combined with Apatinib 、XELOX 、RFA in the treatment of liver metastases of colorectal cancer
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: radiofrequency ablation

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab ：200mg intravenous injection d1 q3w
Drug: Apatinib Mesylate — Apatinib：250mg/d P.O ,qd ,3weeks
Drug: Capecitabine — capecitabine:850mg/m2 P.O ,bid ,d1-d14
Drug: Oxaliplatin — oxaliplatin:130mg/m2 intravenous injection d1 q3w
Radiation: radiofrequency ablation — radiofrequency ablation:between first cycle and second cycle percutaneous

SUMMARY:
To evaluate the safety of karillizumab combined with apatinib mesylate, XELOX and radiofrequency ablation

DETAILED DESCRIPTION:
To evaluate the safety of karillizumab combined with apatinib mesylate, XELOX and radiofrequency ablation.

The 23 patients were enrolled in a 3-week regimen with 200mg Camrelizumab given intravenously every 3weeks and 250mg apatinib mesylate qd ，and 850mg/m2 capecitabine d1-14 and 130mg/m2 oxaliplatin given intravenously d1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Confirmed by pathology (including histology or cytology) as metastatic colorectal adenocarcinoma of the liver (no other metastatic sites)
* Confirmed by CT/MRI/PET - CT/ultrasound examination of liver metastases, the liver metastases number 3 or higher, and the multidisciplinary team (MDT) confirmed for unresectable liver metastases;
* Patients with at least one evaluable or measurable lesions as per RECIST version 1.1 （CT scan length and diameter of tumor lesion≥10mm，CT scan of lymph node lesion was short diameter≥15mm，scan slice thickness 5mm；）
* ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-2 scores
* The expected survival time is more than 3 months
* The main organ function is normal, which should meet the following criteria:

  (1) blood routine examination standards should be met（no blood transfusion within 14 days）

  a．HB≥ 90g/L b. WBC≥3×109/L c. ANC≥1.5×109/L d. PLT≥100×109/L （2）biochemical examination shall comply with the following criteria：
  1. BIL<1.5 normal upper limit ULN
  2. ALT and AST≤5 ULN
  3. Cr≤1.5 ULN，CCR（creatinine clearance rate）≥50ml/min(Cockcroft-Gault formula)
* Women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test。
* Participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.
* Any other malignancy was diagnosed within the first 5 years of the study, except locally treatable and cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast duct, and papillary carcinoma of the thyroid.
* Patients who had received anti-tumor therapy, including chemotherapy, radiotherapy, surgery, endocrine therapy, biological therapy, tumor embolization, targeted therapy and immunotherapy (pd-1 / pd-l1 antibody, anti-pd-l2 antibody, anti-cd137 antibody, ctla-4 antibody, or other drugs/antibodies acting on T cell co-stimulation or checkpoint pathway) within 28 days before enrollment.
* Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; obstruction of the digestive tract with severe infection.
* Distant metastases to sites other than the liver.
* The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)
* Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and unresected gastric primary tumor; patients with the risk of bleeding should take the gastroscopy test, if it is the gastric cancer, and researchers believe that may results in massive digestive tract hemorrhage；coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency
* pregnant or lactating women
* A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation
* Presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia)
* Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g)
* Patients with a history of cardiovascular and cerebrovascular diseases who are still taking oral thrombolytic drugs or anticoagulant drugs
* Patients with uncontrolled epilepsy, central nervous system disease, or mental disorders whose clinical severity, as determined by the investigator, may prevent the signing of the informed consent or have multiple factors that affect oral medications (such as inability to swallow, persistent uncontrolled nausea and vomiting, chronic diarrhea, and intestinal obstruction)
* A person who has previously been allergic to any component of camrilizumab or to any component of the drug under study
* Patients who participate in other clinical studies before or during treatment
* The researchers consider those who were not suitable for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 6 months
  The surgical procedure was total or subtotal proctectomy and hepatectomy with 4 cycles after Conversion therapy

SECONDARY OUTCOMES:
Objective response rate | 6 months
  Objective response rate according to Response Evaluation Criteria in Solid Tumours(RECIST)1.1
pathologic complete response | 6 months
  pathologic complete response (pCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Xiamen University, Xiamen, Fujian, China